CLINICAL TRIAL: NCT00997100
Title: An Exploratory Study to Evaluate Changes in Disease Activity and Biomarkers During Treatment With ABR-215757 in Patients With Mild Active Systemic Lupus Erythematosus (SLE)
Brief Title: Exploratory Study of Changes in Disease Activity and Biomarkers With ABR-215757 in Patients With Mild Active Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09575704; 2009-011245-55 (EudraCT Number)
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus (SLE); ABR-215757; Change in Biomarkers
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — paquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABR-215757 (Other)
  Interventions: Drug: paquinimod (ABR-215757)

INTERVENTIONS:
Drug: paquinimod (ABR-215757) — The initial daily dose of ABR-215757 is changed to 1.5 mg/day. There will be an option to increase the dose to 3.0 mg/day following 28 days of treatment
  Other Names: ABR-215757; paquinimod

SUMMARY:
This is an exploratory open label single arm study to evaluate changes in disease activity and biomarkers in patients with mild active SLE, during treatment with ABR-215757 given as add-on to standard therapy. To be eligible for the study SLE patients should present with symptoms from skin, mouth and/or joints. After a screening period of one week patients will be treated with ABR-215757 for 12 weeks. The initial dose of ABR-215757 will be 1.5 mg/day. There will be an option to increase the dose to 3.0 mg/day following 28 days of treatment. Follow-up visits will take place 4 weeks and 8 weeks after last day of treatment. Disease activity during treatment will be studied using the Systemic Lupus Erythematosus disease Activity Index (SLEDAI-2K) as well as organ system specific disease activity indexes (CLASI for skin involvement and number of swollen/tender joints using 28- and 66/68-joint counts). At specified time points during the study, blood samples and biopsies will be collected for analysis of established and exploratory biomarkers of SLE. Concomitant SLE treatment allowed include: prednisolone or equivalent at a dose of ≤15 mg/day, hydroxychloroquine, azathioprine, methotrexate and mycophenolate mofetil, all at stable doses from specified timepoints prior to the study and throughout the study.

DETAILED DESCRIPTION:
All patients will initially receive ABR-215757 at 1.5 mg/day. There will be an option to increase the dose to 3.0 mg/day following 28 days of treatment. The selected dose levels (1.5 and 3.0 mg/day ABR-215757) are predicted to be effective based on preclinical studies of autoimmune disease including the SLE MRL model. Previous experience in humans as well as in preclinical models supports safe administration of ABR-215757 at doses up to and including 3.0 mg/day. The duration of the study is expected to be sufficient to detect changes in disease activity in this group of patients. Near steady state plasma levels of ABR-215757 in humans are reached in 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at the time of signing the informed consent form
2. Fulfil at least 4 criteria for SLE as defined by the American College of Rheumatology (ACR)
3. Present with active SLE disease with at least one of the following symptoms:

   i) Arthritis - > 2 joints with pain and signs of inflammation (i.e. tenderness, swelling, or effusion) ii) Inflammatory-type skin rash iii) Oral ulcers
4. Laboratory values as follows

   * Hemoglobin ≥ 100 g/L
   * Absolute neutrophil count ≥ 1.0 x 109/L
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * AST (SGOT) / ALT (SGPT) ≤ 2.5 x ULN
5. Ability to take and retain oral medication
6. Ability to sign and date a written informed consent prior to entering the study
7. Willingness and ability to comply with the protocol for the duration of the study

Exclusion Criteria:

1. Active severe SLE flare with central nervous system (CNS) manifestations, active renal lupus, systemic vasculitis, active pericarditis, active pleuritis, active peritonitis or other SLE manifestations requiring treatment not allowed by the study protocol.
2. Severe renal impairment (estimated or measured GFR <50%)
3. Oral treatment with corticosteroids (>15 mg/day prednisolone or equivalent) or changes in corticosteroid dosing within 30 days prior to the first dose of study medication. This also includes intraarticular steroid injections or topical treatment for SLE symptoms. Inhaled or topical steroids may be given for reasons other than SLE disease activity (such as asthma, contact dermatitis) as clinically indicated.
4. Intravenous corticosteroids within 3 months prior to the first dose of study medication.
5. Intravenous cyclophosphamide within 6 months prior to the first dose of study medication.
6. Treatment with anti-rheumatic/immunosuppressive drugs within 3 months prior to first dose of study medication, other than the following medications at stable doses: methotrexate (≤25 mg/week), azathioprine (≤2.5 mg/kg/day), hydroxychloroquine and mycophenolate mofetil (≤3000 mg/day).
7. B-cell depletion therapy (such as treatment with Rituximab) within 12 months prior to the first dose of study medication.
8. Potent inhibitors or inducers of CYP3A4 intravenously or orally within 14 days prior to first dose of study medication.
9. History of myocardial infarction or current uncontrolled angina, severe uncontrolled ventricular arrhythmias, symptomatic congestive heart failure, unstable angina pectoris, or electrocardiographic evidence of acute ischemia.
10. Marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval >450 milliseconds
11. History of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome)
12. Treatment with concomitant medications that prolong the QT interval.
13. History of, or current, ischemic CNS disease.
14. Current malignancy. A 5-year cancer-free period is required with the exception of skin basal or squamous cell carcinoma or cervical cancer in situ that has been excised.
15. Current severe infection
16. Positive result on screening for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV) antibodies.
17. Drug abuse.
18. Major surgery within 3 weeks prior to study entry.
19. Known or suspected hypersensitivity to ABR-215757 or excipients.
20. Female subject of child-bearing potential who is not using a medically accepted safe method of contraception. All female subjects of child-bearing potential must have a negative urine pregnancy test at the Screening and Baseline Visits. As interaction studies between ABR-215757 and oral contraceptives have not yet been performed, women using the contraceptive pill must also use a complementary contraceptive device, i.e. barrier method, during the treatment period and for at least 1 month thereafter.
21. Female subject of child-bearing potential who is pregnant or lactating.
22. Simultaneous participation or participation within 4 months or 5 half lives (whichever is longer) prior to study entry in any other study involving investigational drugs or other experimental therapy.
23. Other significant, unstable medical disease not related to SLE that in the investigator's opinion would confound the study result or put the patient at risk.
24. Patients likely to receive oral or intravenous steroids or immunosuppressant for other non-SLE condition during the study duration, as this will confound the study result.
25. Vaccination within 4 weeks prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in disease activity and biomarkers in patients with mild active SLE treated with ABR-215757 | Patients will be treated for 12 weeks with ABR-215757. During treatment there will be scheduled visits on days 14, 28, 56 and 84. Follow-up visits will take place 29 days and 57 days after last dose of ABR-215757

SECONDARY OUTCOMES:
To assess the safety and tolerability of ABR-215757 in SLE patients with mild active disease. To assess plasma levels of ABR-215757 during the study | Patients will be treated for 12 weeks with ABR-215757. During treatment there will be scheduled visits on days 14, 28, 56 and 84. Follow-up visits will take place 29 days and 57 days after last dose of ABR-215757

CONTACTS AND LOCATIONS:
Overall Officials: Marie Wallén Öhman, Ph.D., Study Director — Active Biotech AB
Locations (4):
- Soren Jacobsen, Copenhagen, Copenhagen, Denmark
- Sweden (3):
  - Dept of Rheumatology, University Hospital in Lund, Lund, Lund
  - Iva Gunnarsson M.D., Stockholm, Stockholm County
  - Lars Rönnblom M.D., Uppsala, Uppsala County